CLINICAL TRIAL: NCT03678636
Title: Clinical and Economic Effectiveness of Testing Chronic Wounds for BPA (Bacterial Protease Activity) Using WOUNDCHEK Bacterial Status: A Pragmatic Randomised Clinical Trial
Brief Title: WOUNDCHEK Bacterial Status Benefits Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woundchek Laboratories BV (Industry)
Collaborators: Pennine Care NHS Foundation Trust (Other Government); Innovate UK (Other Government); Greater Manchester Academic Health Science Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WCL#CT/2018/001
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Intervention Model Description: 100 patients positive for BPA will be randomized to intervention or control treatment. It is anticipated approximately 200-250 patients will be tested assuming a prevalence of BPA of 40-50%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The wound will be treated with a silver antimicrobial dressing appropriate for the exudate level as per manufacturer instructions for use for 2 weeks +/- 3 days, in addition to any necessary standard care (e.g. compression for a venous leg wound).
  Interventions: Device: Silver antimicrobial dressing
- Control (Active Comparator): The wound will be treated as per usual care.
  Interventions: Device: Standard care

INTERVENTIONS:
Device: Silver antimicrobial dressing — Silver dressing suitable for exudate level
  Arms: Intervention
Device: Standard care — Usual care for wound type and condition
  Arms: Control

SUMMARY:
100 chronic wounds asymptomatic for infection that test positive for bacterial protease activity (BPA) on initial screening (approx 250 wounds in total to be tested) will be randomized to intervention or control. 50 patients will receive intervention (silver antimicrobial dressing) in addition to standard care and 50 will receive standard care only (control). Wound healing at 12 weeks will be compared in addition to costs, patient quality of life, referrals to secondary care, surgical interventions, rates of infection and antibiotic use.

DETAILED DESCRIPTION:
A prospective, open randomized controlled study in the community setting. Study participants will be selected from chronic wound patients being treated in the community by Pennine Care NHS Foundation Trust that are not considered to be infected and are not currently being treated with a topical antiseptic dressing. Patients diagnosed with a chronic wound and determined to meet the study inclusion criteria can be enrolled after informed consent. Only one wound is allowed per patient (defined as the 'index wound). If a patient has multiple wounds, the largest wound will be selected.

Enrolled patients will be tested for BPA using the WOUNDCHEK™ Bacterial Status. Patients with negative results will take no further part in the study. Patients with positive results, will be randomized into either the Intervention or the Control arm of the study.

The study aims to enrol 100 patients that test positive for BPA. An expected prevalence of between 40 and 50 percent BPA positive means that between approximately 200 and 250 patients will need to be enrolled and screened to reach the target number of 100 BPA positive wounds.

A total of up to 100 patients with a chronic wound that test positive for BPA during screening will be randomized to receive either a silver antimicrobial dressing appropriate for the wound exudate level for 2 weeks +/- 3 days, in addition to any other standard care requirements (e.g. compression) (Intervention arm) or receive standard care only (Control arm).

The patients will be followed up at 12 weeks post enrolment or within two weeks of wound closure (whichever is earliest). The Research Nurse will visit the patient to measure the wound size or determine if the wound has healed and complete the EQ5D-5L questionnaire.

The initial contact, enrolment and initial test visit for both groups, follow-up visit for both groups, will be conducted by the dedicated Research Nurse. All other patient care will be delivered by the Clinicians from the Community Service.

Data recorded at week 0 (first patient visit for both Control and Intervention groups);

* Eligibility review
* Informed Consent
* WOUNDCHEKTM Bacterial Status result

  • Participants who pass screening (i.e. return a positive BPA result) will be enrolled into the study:
* Randomisation group (if BPA positive)
* Wound type and location
* Wound size (length, width and depth dimensions in cm, +/- 0.1cm)
* Wound age in months
* Wound condition**
* Current treatment
* EQ5D-5L questionnaire

  * Wound condition: Ulcer stage/grade, Tissue Present, Amount and viscosity/colour of exudate, Odour, Surrounding Skin, Pain at wound site.

Data recorded when the wound has healed or at week 12 post randomisation (whichever is soonest) for both Control and Intervention groups;

* EQ5D-5L
* Wound size
* Wound condition (as per the PCFT wound assessment form)
* If healed, what date it healed.
* All visits and treatments by community services clinician in previous 12 weeks
* Episodes of wound infection
* Antibiotic prescriptions related to wound infection
* Any GP consultations or A&E visits associated with the wound.
* Any referrals for treatment in secondary care associated with the wound including any surgical intervention

The study will be expected to last for a year or until completion of the last visit of the 100th patient.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Competence with English language
* Subject has a chronic wound (venous, arterial and mixed etiology leg ulcers, diabetic foot ulcers and pressure ulcers), >1cm2 area which is not showing symptoms of infection or spreading cellulitis / lymphadenitis / lymphangitis and is not receiving treatment for local or systemic infection due to the wound.
* Subject is 18 years of age or older.
* Women must be of non-childbearing potential.
* The wound is more than 4 weeks old.

Exclusion Criteria:

* Women who are pregnant/planning a pregnancy or breastfeeding
* The wound area is ≤1cm2.
* The wound is obviously infected as defined by the Pennine Care Wound Management Formulary or is receiving treatment for local or systemic infection.
* The wound has been diagnosed as being malignant.
* Subject has hypersensitivity of the wound or painful wound surface which prevents touching / swabbing of the wound surface.
* Subject has known allergy to silver dressings.
* Subject is confirmed to be positive for HIV or hepatitis A, B or C.
* Subject is pregnant and/or breastfeeding.
* Subject is unable or unwilling to provide informed consent.
* The wound is related to intravenous drug misuse.
* A designated wound area may only be enrolled once in the study. For example, if an enrolled wound heals to complete closure and then re-opens, it cannot be re-enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Mean wound area percent change | 12 weeks
  To determine whether the use of WOUNDCHEK™ Bacterial Status to guide further management in chronic wounds improves the mean wound area reduction compared to usual care.

SECONDARY OUTCOMES:
Proportion of wounds healed | 12 weeks
  Compare the proportion of wounds healed between study arms
Mean time to healing | 12 weeks
  Compare mean time to healing between study arms.
Total cost of care | 12 weeks
  Aggregate cost of care including dressings, nurse visits and secondary care episodes due to the wound.
Wound infections and antibiotic use | 12 weeks
  Compare the number of wound infections and amount of antibiotic prescribing.
Quality of life using EuroQol EQ-5D-5L | 12 weeks
  EuroQoL EQ-5D-5L is a self-administered questionnaire comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels:1 = no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5 = extreme problems. A unique health state is defined by combining 1 level from each of the 5 dimensions to create a 5 digit code.
Quality of life using EuroQol EQ VAS | 12 weeks
  EuroQoL EQ VAS records the patient's self-rated health on the day of self-reporting on a vertical visual analogue scale from 0 (labelled 'The worst health you can imagine') to 100 (labelled 'The best health you can imagine'). The subscales and EQ VAS will be reported as individual dimensions in order to present any changes in the patient self-report of these health states before and after the intervention.
Referral to secondary care and surgical intervention | 12 weeks
  Compare the number of patients referred to secondary care and having surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Baines, BSc, Principal Investigator — Pennine Care NHS Foundation Trust
Locations (1):
- Pennine Care NHS Foundation Trust, Bury, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available.